CLINICAL TRIAL: NCT03812640
Title: Comparison Between Nylon and Polyglactin Corneal Suture in Pediatric Cataract Surgery: a Randomized Controlled Clinical Trial
Brief Title: Nylon Verus Polyglactin Corneal Suture in Pediatric Cataract Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Mathias Violante Mélega, MD, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Vicryl Unicamp
Record Dates: First submitted 2019-01-18; First posted 2019-01-23 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Endophthalmitis; Cataracts Infantile; Suture, Complication
Keywords: pediatric; cataract; suture; poliglactin; nylon
MeSH Terms: conditions — Endophthalmitis; Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vicryl (Experimental): Vicryl suture
  Interventions: Device: Vicryl suture
- Nylon (Active Comparator): Nylon suture
  Interventions: Device: Nylon suture

INTERVENTIONS:
Device: Vicryl suture — Corneal suture with Vicryl suture
  Arms: Vicryl
Device: Nylon suture — Corneal suture with Nylon suture
  Arms: Nylon

SUMMARY:
Pediatric cataract surgery requires the suturing of the corneal incision in order to maintain the integrity of the eyeball and to help avoid the trauma often caused by scratching in the postoperative period of pediatric surgeries. Traditionally, this suturing is performed using 10-0 nylon material. Because this material is non-absorbable, it must be removed under sedation in cases of complications such as suture loosening, late suture lysis, accumulation of secretion on the suture, corneal neovascularization, and corneal ulceration. The objetive of this study is to compare the rate of postoperative complications and the need for suture removal after pediatric cataract surgery in cases in which nylon (non-absorbable) sutures are used versus cases in which polyglactin (absorbable) sutures are used.

This is a controlled, randomized, prospective, single-center study performed on patients undergoing pediatric cataract surgery at the Clinical Hospital of the University of Campinas (UNICAMP). The volunteers for whom cataract extraction surgery has been indicated and who have signed the ICF (or whose ICF has been signed by a parent or guardian) will undergo cataract surgery and the cornea will be sutured using a polyglactin 910 suture (Vicryl® 10-0). In the control group (Group B), the cornea will be sutured using nylon 10-0 sutures (the current routine procedure). All patients will be monitored for six months and will receive complete ophthalmological evaluations in order to determine whether they experience any suture-related complications and whether sutures must be removed under sedation. A lower incidence of complications and a less frequent need for suture removal under sedation are expected in the group receiving Vicryl® sutures.

DETAILED DESCRIPTION:
Patients who are diagnosed with cataracts and for whom surgery is indicated shall be evaluated (as much as possible based on their ability to cooperate with the assessment) in terms of their visual acuity and refractive error via biomicroscopy, automated keratometry (Auto Kerato Refractometer KR 8000® Alcon), Goldmann applanation tonometry, fundoscopy, and biometric assessment (Ocuscan RxP® Alcon or Lenstar LS900® Haag-Streit International).

Patients who choose to sign (or whose guardians choose to sign) the informed consent form after being informed of all of the aspects of the surgery and this trial shall be randomly divided into one of two groups that shall be approximately equal in size and stratified by age.

* Up to 6 months of age
* From 6 to 12 months of age
* From 1 to 3 years of age
* From 3 to 6 years of age
* Older than 6 years Patients in Group A will have their surgical incisions sutured with polyglactin 10-0 material (Vicryl®, composed of polyglactin 910, 10-0 diameter, absorbable, a 0.62 cm, 3/8 circle needle) at the end of cataract surgery followed by the use of 0.5% moxifloxacin and 0.1% dexamethasone eye drops before the bandage is applied. Patients in Group B will have their surgical incisions sutured with nylon 10-0 material (Vicryl®, composed of nylon monofilament, 10-0 diameter, absorbable, a 0.55 cm, 1/2 circle needle) at the end of cataract surgery followed by the use of 0.5% moxifloxacin and 0.1% dexamethasone eye drops before the bandage is applied.

Cataract surgery will be performed using the standardized protocol in the Ophthalmology department of UNICAMP by fourth-year ophthalmology residents with experience in pediatric cataract surgery. Preoperative pupil dilation shall be performed through the use of 2.5% phenylephrine and 1% tropicamide 3 times in five-minute increments. General anesthesia shall be performed. Skin sterilization shall be performed using an aqueous solution of 10% povidone-iodine. After the sterile surgical field is established and the eyelashes are isolated, 4 eye drops containing 5% povidone-iodine shall be administered in the conjunctival sac with subsequent irrigation using a 10% balanced salt solution. In cases of allergy to povidone-iodine, an aqueous solution of 0.05% chlorhexidine shall be used. The main incision (either a clear corneal incision or a scleral tunnel) will be 2.2 mm to 3.0 mm, and aspiration will be applied using the Infiniti® or Laureate® phacoemulsifier (Alcon) with a foldable AcrySof® intraocular lens (Alcon) and a posterior capsulotomy with an automated vitrectomy only in cases in which it is indicated.

Neither patients nor surgeons will be masked to the study treatment. The postoperative consultations will be held on the first, seventh, thirtieth, ninetieth, one hundred and twentieth, and one hundred and eightieth postoperative days and will include visual acuity assessments, refractive error assessments, keratometry , biomicroscopy, applanation tonometry, and fundoscopy, depending on the patient's age and ability to cooperate. If a necessary exam is not possible in a clinical setting, it will be performed under sedation in the surgical center.

Primary outcome: frequency of complications associated with sutures in each group.

Secondary outcome: need for suture removal under sedation in each group. The following will be defined as suture-related complications: corneal neovascularization close to the suture, loosening of the suture, accumulation of mucus on the suture, early rupture (within 2 weeks or less) of the suture, aqueous humor leakage through the incision (as determined by the Seidel test), prolapse of the iris through the incision site, infectious or traumatic keratitis, endophthalmitis and giant papillary conjunctivitis as observed in a biomicroscopy exam using a slit lamp.

Based on the frequency of suture-related complications described in the literature and using a two-tailed 95% confidence interval, 80% power, an exposed/unexposed radius of 1, and a null frequency of complications in the polyglactin suture group, approximately 40 subjects are needed for each group. UNICAMP performs an average of 75 pediatric cataract surgeries per year. Thus, there is a perspective for patient inclusion and study completion of just over one year.

ELIGIBILITY:
Inclusion Criteria:

* Patients up to 14 years of age who are clinically qualified to undergo pediatric cataract surgery

Exclusion Criteria:

* Traumatic cataract with ocular perforation
* Cataract surgery associated with other procedures, such as glaucoma filtering surgery, vitreoretinal surgery, and cornea surgery
* Signs of ocular or periocular infection
* Advanced glaucoma

Ages: 30 Days to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-09-01 (Estimated); Study Completion 2019-10-01 (Estimated)

PRIMARY OUTCOMES:
frequency of complications associated with sutures in each group | 180 days
  frequency of complications associated with sutures in each group

SECONDARY OUTCOMES:
need for suture removal under sedation in each group. | 180 days
  need for suture removal under sedation in each group.

CONTACTS AND LOCATIONS:
Locations (1):
- Mathias Violante Mélega, Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Foster A, Gilbert C, Rahi J. Epidemiology of cataract in childhood: a global perspective. J Cataract Refract Surg. 1997;23 Suppl 1:601-4. doi: 10.1016/s0886-3350(97)80040-5. PMID 9278811
- [Background] Gilbert CE, Wood M, Waddel K, Foster A. Causes of childhood blindness in east Africa: results in 491 pupils attending 17 schools for the blind in Malawi, Kenya and Uganda. Ophthalmic Epidemiol. 1995 Jun;2(2):77-84. doi: 10.3109/09286589509057086. PMID 7585238
- [Background] Haargaard B, Wohlfahrt J, Fledelius HC, Rosenberg T, Melbye M. Incidence and cumulative risk of childhood cataract in a cohort of 2.6 million Danish children. Invest Ophthalmol Vis Sci. 2004 May;45(5):1316-20. doi: 10.1167/iovs.03-0635. PMID 15111583
- [Background] WHO | Priority eye diseases. WHO [Internet]. 2014 [cited 2017 Dec 29]; Available from: http://www.who.int/blindness/causes/priority/en/index3.html
- [Background] Wilson BME. Pediatric Cataracts : Overview Classification ( Categorization ). 2016;
- [Background] Heaven CJ, Boase DL. Suppurative keratitis with endophthalmitis due to biodegraded full thickness monofilament nylon corneal sutures. Eur J Implant Refract Surg [Internet]. 1993;5(3):164-8. Available from: http://dx.doi.org/10.1016/S0955-3681(13)80436-4
- [Background] Lee BJ, Smith SD, Jeng BH. Suture-related corneal infections after clear corneal cataract surgery. J Cataract Refract Surg. 2009 May;35(5):939-42. doi: 10.1016/j.jcrs.2008.10.061. PMID 19393897
- [Background] Culbert RB, Devenyi RG. Bacterial endophthalmitis after suture removal. J Cataract Refract Surg. 1999 May;25(5):725-7. doi: 10.1016/s0886-3350(99)00020-6. PMID 10330655
- [Background] Khurshid GS, Fahy GT. Endophthalmitis secondary to corneal sutures: series of delayed-onset keratitis requiring intravitreal antibiotics. J Cataract Refract Surg. 2003 Jul;29(7):1370-2. doi: 10.1016/s0886-3350(03)00404-8. PMID 12900247
- [Background] Acheson JF, Lyons CJ. Ocular morbidity due to monofilament nylon corneal sutures. Eye (Lond). 1991;5 ( Pt 1):106-12. doi: 10.1038/eye.1991.20. No abstract available. PMID 2060657
- [Background] Danjoux JP, Reck AC. Corneal sutures: is routine removal really necessary? Eye (Lond). 1994;8 ( Pt 3):339-42. doi: 10.1038/eye.1994.70. PMID 7958043
- [Background] Bainbridge JW, Teimory M, Kirwan JF, Rostron CK. A prospective controlled study of a 10/0 absorbable polyglactin suture for corneal incision phacoemulsification. Eye (Lond). 1998;12 ( Pt 3a):399-402. doi: 10.1038/eye.1998.94. PMID 9775239
- [Background] Bar-Sela SM, Spierer O, Spierer A. Suture-related complications after congenital cataract surgery: Vicryl versus Mersilene sutures. J Cataract Refract Surg. 2007 Feb;33(2):301-4. doi: 10.1016/j.jcrs.2006.10.039. PMID 17276274
- [Derived] Melega MV, Dos Reis R, Lira RPC, de Oliveira DF, Arieta CEL, Alves M. Comparison Between Nylon and Polyglactin Sutures in Pediatric Cataract Surgery: A Randomized Controlled Clinical Trial. Front Med (Lausanne). 2021 Aug 27;8:700793. doi: 10.3389/fmed.2021.700793. eCollection 2021. PMID 34513873